CLINICAL TRIAL: NCT02533791
Title: Safety and Immunogenicity of a Booster Dose of the Recombinant Ebola Adenovirus Vector Vaccine (Ad5-EBOV) in Healthy Adults After Primary Immunization
Brief Title: A Booster Dose of Ad5-EBOV in Healthy Adults After Primary Immunization
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Beijing Institute of Biotechnology (Other); Tianjin Cansino Biotechnology Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JSVCT020-2
Record Dates: First submitted 2015-08-21; First posted 2015-08-27 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Ebola Virus Disease
Keywords: Safety; immunogenicity; Ebola vaccine; boosting
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- low dose group (Experimental): 4×10^10vp/1ml Ebola Zaire vaccine (Ad5-EBOV)
  Interventions: Biological: 4×10^10vp/1ml Ebola Zaire vaccine (Ad5-EBOV)
- high dose group (Experimental): 1.6×10^11vp/2ml Ebola Zaire vaccine (Ad5-EBOV)
  Interventions: Biological: 1.6×10^11vp/2ml Ebola Zaire vaccine (Ad5-EBOV)
- placebo group (Placebo Comparator): placebo
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: 4×10^10vp/1ml Ebola Zaire vaccine (Ad5-EBOV) — one dose, 4×10^10vp/1ml per dose
  Arms: low dose group
Biological: 1.6×10^11vp/2ml Ebola Zaire vaccine (Ad5-EBOV) — two doses, 0.8×10^11vp/1ml per dose, with one dose to each arm at the same time
  Arms: high dose group
Biological: placebo
  Arms: placebo group

SUMMARY:
Since its first outbreak occurred in 1976, Zaire Ebola virus have been associated with 14 outbreaks reported up to 2014. The Zaire Ebola virus in 2014 causing the most serious outbreak was considered to be a new epidemic strain, with GP homology of the gene was only 97.6%, compared to the GP gene of the strain in 1976. This investigational Ad5-EBOV vaccine was developed according to the 2014 epidemic Zaire strain and formulated as freeze-dry products which could be stored at 4℃.

In 2014, a single center, double-blind, placebo control, dose-escalation phase 1 clinical trial was performed in Taizhou, China. Our findings show that the Ad5-EBOV vaccine is safe and robustly immunogenic. One shot of the high dose vaccine could mount glycoprotein-specific humoral and T-cell response against Ebola virus in 14 days. The investigators intent to evaluate the safety and immunogenicity of a booster dose of the recombinant Ebola adenovirus vector vaccine (Ad5-EBOV) in healthy adults after primary immunization in this add in study. The investigators expect that the boosting immunization with a same vaccine for primary immunization is possible and could confer a longer-lived protection when needed.

The phase I trial has been unblind 28 days after the primary vaccination, but all the subjects are still kept blind as well as the laboratory staffs. Therefore, this booster vaccination trial will be conduct in single blind.

ELIGIBILITY:
Inclusion Criteria:

* Participants who enrolled in the initial study, and completed the primary vaccination.
* Able to understand the content of the additional informed consent and willing to sign the additional informed consent for the boosting study
* Able and willing to complete a one-month follow-up.
* HIV negative
* Axillary temperature ≤37.0°C on the day of enrollment
* General good health as established by medical history and physical examination.

Exclusion Criteria:

New occurrence of any of the following situation after the primary vaccination:

* Subject that has a medical history of any of the following: allergic history of any vaccination or drugs, or allergic to any ingredient of the Ad5-EBOV vaccine, such as mannitol
* Woman who become pregnant after the primary vaccination or is positive in β-HCG (human chorionic gonadotropin) pregnancy test (urine) on day of enrollment for the boosting study
* Any acute fever disease or infections in last 7 days
* Not well-controlled chronic illness, such as asthma, diabetes, or thyroid disease
* Hereditary angioneurotic edema or acquired angioneurotic edema
* Urticaria in last 6 months
* Asplenia or functional asplenia
* Platelet disorder or other bleeding disorder may cause injection contraindication
* Faint at the sight of blood or needles.
* Prior administration of immunodepressant or corticosteroids, antianaphylaxis treatment, cytotoxic treatment in last 6 months
* Prior administration of blood products in last 4 months
* Prior administration of other research medicines in last 1 month
* Prior administration of attenuated vaccine in last 1 month
* Prior administration of inactivated vaccine in last 14 days
* Current anti-tuberculosis prophylaxis or therapy
* Any condition that in the opinion of the investigators may interfere with the evaluation of study objectives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse reactions after vaccination | within 7 days after the boosting
  Occurrence of adverse reactions within 7 days after vaccination with the Ebola Zaire vaccine (Ad5-EBOV)
Specific anti-EBOV antibody responses to the Ebola Zaire vaccine (Ad5-EBOV) | 28 days after the boosting
  Specific anti-EBOV antibody responses to the Ebola Zaire vaccine (Ad5-EBOV) as measured by ELISA
Specific T cell immune responses to the Ebola Zaire vaccine (Ad5-EBOV) | 28 days after the boosting
  Specific T cell immune responses to the Ebola Zaire vaccine (Ad5-EBOV)

SECONDARY OUTCOMES:
Occurrence of adverse events after the vaccination | within 28 days after the boosting
  Occurrence of adverse events within 28 days after vaccination with the Ebola Zaire vaccine (Ad5-EBOV)
Occurrence of serious adverse events after the vaccination | within 28 days after the boosting
  Occurrence of serious adverse events within 28 days after the vaccination with the Ebola Zaire vaccine (Ad5-EBOV)
Serum neutralizing antibody against the Ad5-vector | 28 days after the boosting
  Serum neutralizing antibody against the Ad5-vector 28 days after the boosting

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Cai Zhu, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Phase 1 vaccine clinical trial center of Jiangsu Provincial Center for Disease Control and Prevention, Taizhou, Jiangsu, China

REFERENCES:
- [Derived] Li JX, Hou LH, Meng FY, Wu SP, Hu YM, Liang Q, Chu K, Zhang Z, Xu JJ, Tang R, Wang WJ, Liu P, Hu JL, Luo L, Jiang R, Zhu FC, Chen W. Immunity duration of a recombinant adenovirus type-5 vector-based Ebola vaccine and a homologous prime-boost immunisation in healthy adults in China: final report of a randomised, double-blind, placebo-controlled, phase 1 trial. Lancet Glob Health. 2017 Mar;5(3):e324-e334. doi: 10.1016/S2214-109X(16)30367-9. Epub 2016 Dec 23. PMID 28017642